CLINICAL TRIAL: NCT07172750
Title: The Effect of Education on Patients' Attitudes Towards Preventing Catheter-Associated Urinary Tract Infections and Anxiety After Urologic Surgery
Brief Title: The Effect of Education on Patients' Attitudes and Anxiety Towards CAUTI Prevention
Acronym: CAUTI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kübra ATA, MSc canditate of nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulUC-KATA
Record Dates: First submitted 2025-08-28; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Catheter Associated Urinary Tract Infection; Indwelling Urinary Catheter; Urologic Surgery
Keywords: Catheter associated urinary tract infection; Anxiety; self-care; Urologic Surgery; patient education
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group: Urinary catheter care training (Experimental): Urology patients in this group will receive urinary catheter care training based on Roper, Logan, Tierney Model of Nursing (based on Activities of Living).
  Interventions: Other: Education on Urinary Catheter Care
- No Intervention: Control Group: Standard discharge training (No Intervention): Urology patients in this group will not receive any training other than the discharge training routinely applied in the clinic.

INTERVENTIONS:
Other: Education on Urinary Catheter Care — Urinary catheter care training based on the Roper, Logan, and Tierney Lifestyle Model was developed based on daily living activities.
  A training booklet was created based on 11 daily living activities (providing and maintaining a safe environment, communication, breathing, nutrition, etc.).
  To increase the effectiveness of the training, a booklet based on this model will be prepared and used as a guide in the training program.
  Arms: Experimental: Intervention Group: Urinary catheter care training

SUMMARY:
This research will be carried out determine the effect of education given to patients after urological surgery on their attitudes and anxiety levels towards preventing catheter-related urinary tract infections.

DETAILED DESCRIPTION:
Urology surgeries are surgical procedures performed to treat diseases of the kidneys, ureters, bladder, prostate, and urethra. Urinary catheterization is a procedure performed to drain urine from the bladder or collect a urine sample using a catheter. A urinary catheter is inserted in 15-25% of hospitalized patients during their hospital stay, and many patients are discharged home with a urinary catheter after urology surgery.

Urinary tract infection (UTI) is the most common healthcare-associated infection, accounting for 36% of all healthcare-associated infections.

Approximately 75% of hospital-acquired urinary tract infections are associated with urinary catheters. A catheter-associated urinary tract infection is defined as a urinary tract infection that occurs when a urinary catheter has been in place for at least two days. Patients discharged with a urinary catheter; They may encounter various problems, including urinary tract infections, bag emptying, catheter changes, clothing adjustments, (hand) hygiene, odor, and catheter kinking. They may also experience physical and psychosocial difficulties related to catheter care. These problems also bring with them the risk of urinary catheter-related complications. Today, nursing practice prioritizes supporting individuals and families in their own self-care by providing them with the necessary knowledge and skills, rather than assuming full responsibility for their care.

Guidelines for preventing catheter-associated urinary tract infections recommend involving patients and their families in their care to prevent these infections.Therefore, nurses, in their role as educators, should provide training to ensure patients maintain their daily activities with their catheters, particularly regarding catheter care.

In this direction, this study will attempt to reveal the effects of post-urological surgery education on patients' attitudes and anxiety levels towards preventing catheter-related urinary tract infections.

This research will be conducted in a prospective, randomized experimental design with pretest-posttest experimental and control groups. The sample size of the study will consist of urology patients who meet the inclusion criteria and agree to participate in the study.The patients to be included in the sample of the study will be randomly divided into two groups as experimental and control groups. The study sample size was calculated using data from a similar study in the literature using the G*Power 3.1.9.7 program for an independent samples t-test, with a test power (power) of 0.80, a confidence level of 95% (1-α), and an effect size of f=0.64, for a total of 62 patients (31 in the experimental group and 31 in the control group), with a minimum of 31 patients in each group.

However, considering data loss, the plan is to include at least 70 patients (35 in the experimental group and 35 in the control group).

Data will be collected using the "Individual Characteristics Form," the "State and Trait Anxiety Inventory," and the "Attitude Scale for Preventing Catheter-Associated Urinary Tract Infections in Patients with Indwelling Urinary Catheters." The "Patient Education Material Evaluation Tool (HEMDA)" will be used to evaluate the educational materials and will be submitted to an expert for review. R ver. 2.15.3 program (R Core Team, 2013) will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over,
* Male patients,
* Discharged with a urinary catheter after TURP, HOLEP, Internal Urethrotomy, and Open Prostatectomy surgeries at the urology department of the University Hospital where the study will be conducted,
* Possess the cognitive, affective, and psychomotor skills to perform self-care (no coordination problems affecting the upper extremities),
* Are literate,
* Have no visual or auditory communication problems,
* Have no previous psychiatric disorder/diagnosis and are not currently taking medication for psychiatric disorders,
* Individuals who volunteer to participate in the study will be included.

Exclusion Criteria:

* Patients who are under 18 years of age,
* Female patients,
* Patients who have undergone surgeries other than TUR-P, HOLEP, Internal Urethrotomy, and Open Prostatectomy,
* Patients with an oncological diagnosis and ongoing care/treatment, or who have previously received oncological treatment,
* Patients who develop postoperative complications/whose general health deteriorates, who do not wish to participate in the study, or who wish to withdraw/exit from any aspect of the study will not be included in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
CAUTI Prevention Attitude | Time Frame: "Baseline (discharge planning day)" Time Frame: "Day of catheter removal (within 3-7 days after discharge)
  The scale developed by Koçyiğit Kavak et al. (2024) is a 31-item instrument designed to assess patients' attitudes towards preventing catheter-associated urinary tract infections. The Turkish validity and reliability study of the scale was conducted by Koçyiğit Kavak et al. in 2024. The Cronbach's alpha coefficient of the scale was reported as 0.882. The scale consists of 31 items in a five-point Likert type format, with response options ranging from "Never = 1," "Rarely = 2," "Sometimes = 3," "Often = 4," to "Always = 5." The minimum possible score is 31, and the maximum score is 155. Higher scores indicate more positive patient attitudes towards preventing catheter-associated urinary tract infections.
Anxiety | Time Frame: "Baseline (discharge planning day)" Time Frame: "Day of catheter removal (within 3-7 days after discharge)
  To determine individuals' anxiety levels, the State-Trait Anxiety Inventory (STAI) will be used. The scale consists of a total of 40 items and is a four-point Likert-type instrument composed of two subscales: the State Anxiety Inventory (first 20 items) and the Trait Anxiety Inventory (last 20 items). The State Anxiety subscale measures how an individual feels at a particular time and under specific conditions, whereas the Trait Anxiety subscale assesses how an individual generally feels regardless of the situation and conditions. A score between 0-19 indicates no anxiety, 20-39 indicates mild anxiety, 40-59 indicates moderate anxiety, and 60-79 indicates severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin ÖZAKGÜL, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul University-Cerrahpasa, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is conducted as part of a master thesis, and the collected data will be used only for the purposes of the study and related publications

REFERENCES:
- [Background] Safdar N, Codispoti N, Purvis S, Knobloch MJ. Patient perspectives on indwelling urinary catheter use in the hospital. Am J Infect Control. 2016 Mar 1;44(3):e23-4. doi: 10.1016/j.ajic.2015.10.011. Epub 2015 Dec 14. PMID 26698670
- [Background] Inman DM, Jacobson TM, Maxson PM, Wang H, Lohse CM. Effects of urinary catheter education for patients undergoing prostatectomy. Urol Nurs. 2013 Nov-Dec;33(6):289-98. PMID 24592522
- [Background] Drake MJ, Clavica F, Murphy C, Fader MJ. Innovating Indwelling Catheter Design to Counteract Urinary Tract Infection. Eur Urol Focus. 2024 Sep;10(5):713-719. doi: 10.1016/j.euf.2024.09.015. Epub 2024 Sep 28. PMID 39341718
- [Background] Ryan P, Sawin KJ. The Individual and Family Self-Management Theory: background and perspectives on context, process, and outcomes. Nurs Outlook. 2009 Jul-Aug;57(4):217-225.e6. doi: 10.1016/j.outlook.2008.10.004. PMID 19631064
- [Background] Laan BJ, Nieuwkerk PT, Geerlings SE. Patients knowledge and experience with urinary and peripheral intravenous catheters. World J Urol. 2020 Jan;38(1):57-62. doi: 10.1007/s00345-018-02623-4. Epub 2019 Jan 24. PMID 30680418
- [Background] Garcia DM, Makic MBF, Casey K. Rounding and Quick Access Education to Reduce Catheter-Associated Urinary Tract Infections. Clin Nurse Spec. 2023 May-Jun 01;37(3):117-123. doi: 10.1097/NUR.0000000000000741. PMID 37058702
- [Background] Parker V, Giles M, Graham L, Suthers B, Watts W, O'Brien T, Searles A. Avoiding inappropriate urinary catheter use and catheter-associated urinary tract infection (CAUTI): a pre-post control intervention study. BMC Health Serv Res. 2017 May 2;17(1):314. doi: 10.1186/s12913-017-2268-2. PMID 28464815